CLINICAL TRIAL: NCT06653257
Title: Outcomes of a 5-Year Active Surveillance Program in Bethesda IV-VI Thyroid Nodules
Brief Title: Active Surveillance Program in Thyroid Nodules
Status: Not yet recruiting | Type: Observational
Sponsor: Centro de Excelencia en Enfermedades de Cabeza y Cuello (Other)
Collaborators: Hospital Alma Mater de Antioquia (Unknown); Hospital San Vicente Fundación (Other); Clinica Somer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Nodule
Keywords: thyroid; nodule; bethesda; active surveillance
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bethesda IV-VI report: thyroid nodules who underwent FNAC with a Bethesda IV-VI report
  Interventions: Other: Active surveillance

INTERVENTIONS:
Other: Active surveillance — a non-operative management strategy aimed at avoiding unnecessary surgery in patients with thyroid nodules with a cytopathological diagnosis of Bethesda IV-VI, who do not present clinical or imaging characteristics suggesting malignancy and/or aggressiveness.

SUMMARY:
Overview This study focuses on thyroid nodules, specifically the Bethesda IV-VI categories, which have uncertain or suspicious malignancy. The idea is to observe and monitor these nodules instead of opting for immediate surgery, a practice known as active surveillance. The main goal of active surveillance is to avoid unnecessary surgeries, which can lead to complications like nerve damage or hypoparathyroidism.

Problem and Objectives Thyroid nodules in these Bethesda categories can be cancerous, but not all require immediate removal. Active surveillance tracks nodule growth and other changes using regular ultrasounds and clinical checkups. This approach is gaining popularity, especially in Japan, Europe, and the U.S., but there's still a need for more data, particularly in Latin America.

The primary objectives of the study are:

General: To describe the clinical and imaging characteristics of patients with Bethesda IV-VI nodules under active surveillance.

Specific: To measure surgery rates, reasons for surgery, and how long patients can avoid surgery.

Methodology This study is a multicenter historical cohort study, which will look at patients treated from 2019 to 2023 in different hospitals. Patients included in the study are those with Bethesda IV-VI thyroid nodules, who are over 18 and have been managed without immediate thyroid surgery. Data will be collected from medical records and imaging reports, and patients will be followed up to document any changes in their nodules, including growth or metastasis.

Expected Impact The study aims to determine whether active surveillance can safely delay or avoid surgery for selected patients. It could have a significant impact on clinical decision-making, improving patient outcomes and reducing unnecessary surgeries, especially within the Colombian healthcare system. If successful, this approach could reduce costs and improve the quality of life for patients with thyroid nodules.

Ethical Considerations The study will follow ethical guidelines, ensuring patient confidentiality and classifying the research as "no-risk," meaning it involves minimal risk to the participants.

DETAILED DESCRIPTION:
1. Overview Papillary thyroid carcinoma (PTC) is the most common malignant tumor of the thyroid gland. To date, several clinicopathological characteristics have been identified that predict poor prognosis in patients with PTC, including advanced age, extrathyroidal and/or extranodal extension, lymph node metastasis and/or distant metastasis, and tumor size. ¹ Active surveillance in thyroid nodules has been proposed as an alternative to surgery in patients with indeterminate or suspicious nodules for malignancy on fine-needle aspiration cytology (Bethesda IV, V, and VI). Active surveillance involves the systematic and regular observation of nodules through imaging techniques and clinical examination to detect changes in size and ultrasonographic characteristics of the nodules.

   The main advantage of active surveillance is that it can avoid thyroid surgery in selected patients, thereby reducing the rate of surgery-related complications. Several studies have shown that most Bethesda IV-VI thyroid nodules exhibit non-aggressive behavior, and many patients do not require surgery.

   For example, Ito et al.¹ reported that 88% of patients with Bethesda V-VI thyroid nodules who underwent active surveillance did not require surgery during a 5-year follow-up. In addition, active surveillance has been associated with a reduction in the rate of surgery and, consequently, surgery-related complications.2 Another advantage of active surveillance is that it can be a cost-effective alternative compared to surgery. Thyroid surgery is an invasive procedure that can be expensive. On the other hand, it involves regular doctor visits and imaging tests, which are less costly than surgery. In a cost-effectiveness study, active surveillance was associated with a savings of USD $16,542 per patient compared to surgery.3 However, active surveillance also has some limitations and disadvantages. One limitation is that it requires long-term follow-up and a high level of patient compliance to be effective. Patients undergoing active surveillance must be closely monitored for changes in the nodules that may indicate the need for surgery. Additionally, some patients may experience anxiety or stress due to the uncertainty of not knowing whether they have cancer, or if confirmed, not understanding the behavior the cancer will take. 3,4
2. Problem Statement Thyroid nodules with a cytopathological diagnosis of Bethesda IV-VI represent a significant clinical challenge due to the possibility of malignancy and the implications this has for therapeutic management. The current standard recommendation includes thyroidectomy (partial or total); however, these interventions are not without risks and/or morbidity for the patient. Although active surveillance has been proposed as a conservative alternative, especially for nodules with suspicious characteristics and/or nodules with confirmed malignancy that meet certain criteria, there is still a lack of studies in the literature that systematically evaluate its efficacy and safety in our setting.

   Active surveillance aims to avoid overtreatment by identifying and monitoring nodules with high-risk imaging or cytopathological characteristics, allowing for selective surgical intervention only when there is evidence of progression, such as nodule growth or the appearance of lymph node metastases. While preliminary studies on active surveillance in Bethesda V-VI nodules exist, the clinical and ultrasound behavior of patients managed with this strategy has not been sufficiently characterized, nor has its impact on reducing unnecessary surgical procedures been clearly determined. Therefore, a systematic evaluation of the evolution of Bethesda IV-VI thyroid nodules under an active surveillance program is essential.

   This study aims to describe the initial clinical, imaging, and cytopathological characteristics, as well as the documentation of changes during follow-up, including the nodule growth rate, the appearance of lymph node metastases, and the need for conversion to surgery. The evidence generated could guide future clinical management, optimizing the balance between safety and the reduction of unnecessary surgical interventions.

   Research Question In patients with thyroid nodules with a cytopathological diagnosis of Bethesda IV-VI, how do their clinical and imaging status evolve under an active surveillance program, and what factors are associated with the need for conversion to surgery?
3. Marco conceptual Active surveillance in thyroid nodules is a non-operative management strategy aimed at avoiding unnecessary surgery in patients with thyroid nodules with a cytopathological diagnosis of Bethesda IV-VI, who do not present clinical or imaging characteristics suggesting malignancy and/or aggressiveness. The history of active surveillance dates back to the 1990s in Japan, where the first studies were conducted to evaluate the safety of this strategy. Ito et al. were the first to report active surveillance as a safe alternative for managing thyroid nodules with low suspicion of malignancy in Japanese patients. 2 Since then, numerous studies have evaluated the effectiveness and safety of active surveillance in different populations and settings. Sugitani et al.⁵ published a retrospective study of 54 Japanese patients who had undergone active follow-up for an average of 5 years. The study found that 50% of the thyroid nodules had not shown significant changes in size or ultrasound characteristics during follow-up, and none of the patients had developed metastasis or thyroid cancer-related death during the follow-up period.

   In Europe, active surveillance has been more frequently used in patients with small, low-risk thyroid nodules. The European Thyroid Association (ETA) published a clinical guideline recommending active surveillance as an option for managing thyroid nodules smaller than 1 cm with low suspicion of malignancy.⁶ A European study found that active surveillance was safe in the follow-up of low-suspicion thyroid nodules, with a thyroid cancer-related mortality rate of 0.2%.⁷ In the United States, active surveillance has been more frequently used in patients with Bethesda V-VI thyroid nodules. The American Thyroid Association (ATA) issued a statement recognizing active surveillance as a reasonable alternative for the management of low-suspicion thyroid nodules in select patients (Bethesda IV), as well as in thyroid carcinoma (Bethesda V-VI) in small nodules without lymph node involvement.⁸ A retrospective study found that active surveillance was safe and effective in the long-term follow-up of these patients, with a thyroid cancer-related mortality rate of 0.5%.³ In Latin America, studies on active surveillance of thyroid nodules have also been conducted. One of the most important studies was carried out in Colombia by Sanabria.⁹,¹⁰ This study included a total of 109 patients with Bethesda V-VI thyroid nodules who were followed for a period of 36 months. The results showed a growth rate of 21%, with only 6% of the nodules showing growth greater than 50%, and these patients were taken to surgery. García-Lozano and Sanabria described the follow-up of 51 patients with Bethesda IV thyroid nodules, with growth >3 mm in 4 patients (7.84%). The results showed that only 5% of patients undergoing active surveillance required surgery due to nodule growth.¹¹ In Brazil, a prospective study on active surveillance of thyroid nodules with Bethesda V-VI cytology was conducted, where only 1 out of 70 patients showed tumor progression after 30 months of follow-up.¹² Pitoia reported the follow-up of 36 patients diagnosed with thyroid carcinoma, of which 17% showed an increase in tumor size over a period of 4.6 years, with no evidence of lymph node metastasis.¹³ It is important to highlight that thyroid surgery, although curative in many cases, is not without risks. Among the most common complications are hypoparathyroidism and recurrent laryngeal nerve injury, which can cause dysphonia or even severe respiratory problems. Avoiding these complications through active surveillance without affecting the patient's oncological prognosis is an attractive option, especially for selected patients. Based on the literature and the experience from various high-volume centers, active surveillance is a safe alternative to surgical management, leaving surgery as an option only if there are changes in tumor characteristics.
4. Objectives General Objective To describe the clinical and imaging characteristics of a cohort of patients with thyroid nodules and fine-needle aspiration cytology (FNAC) categorized as Bethesda IV-VI, who were managed with active surveillance.

   Specific Objectives
   * To measure the frequency of clinical characteristics in patients (demographics, nodule characteristics, imaging, and pathology in FNAC).
   * To define the incidence of surgery, the reason for surgical intervention, and surgery-free survival.
5. Methodology Design A descriptive, multicenter, historical cohort study. (Participating institutions: HUSVF, HAMA, Center of Excellence in Head and Neck Diseases - CEXCA, Somer Clinic)

Population Patients with thyroid nodules who underwent FNAC with a Bethesda IV-VI report. Inclusion Criteria

1. Patients with thyroid nodules and FNAC with a report corresponding to Bethesda category IV-VI, treated at the following health centers: HUSVF, HAMA, Center of Excellence in Head and Neck Diseases - CEXCA, Somer Clinic.
2. Patients classified as low-risk tumors (intrathyroidal, with no evidence of locoregional or distant metastasis).
3. Patients not subjected to thyroidectomy as the initial treatment.
4. Patients over 18 years of age. Exclusion Criteria

1. Patients with a second head and neck cancer. 2. Patients with clinical or imaging evidence of thyroid malignancy with lymph node or distant metastasis confirmed by pathology.

Sample Selection of consecutive cases of patients who meet the inclusion and exclusion criteria at the hospital from January 2019 to December 2023. Patients treated in the head and neck surgery clinic who presented with thyroid nodules and had FNAC results with Bethesda IV-VI will be selected. Records of ultrasound reports and biopsy pathology results will be taken. A follow-up evaluation will be performed based on subsequent clinical controls with high-resolution ultrasound reports, new biopsies, or indication for surgery.

Data Analysis Data analysis will be conducted using Microsoft Excel for the initial organization of information. A comprehensive descriptive analysis will be performed, covering the clinical, cytopathological, and imaging characteristics of patients undergoing active surveillance. Variables such as age, sex, initial nodule size, ultrasound findings, and cytological results will be considered. For continuous variables, measures of central tendency (mean, median) and dispersion (standard deviation, interquartile ranges) will be calculated to provide a clear understanding of data distribution. Categorical variables will be presented as absolute frequencies and percentages to facilitate interpretation.

For survival analysis, Kaplan-Meier curves will be used to estimate the probability of remaining under active surveillance without significant nodule progression or the need for surgical intervention over time. To identify factors associated with the time to nodule progression or the need for surgery, a Cox proportional hazards model will be applied. This model will assess the relationship between various variables and the risk of progression, providing a multivariate analysis that identifies independent predictors of progression or surgical intervention.

Variables Variable Type of Variable Definition for the Study Sociodemographic Variables Age Quantitative Age in completed years at the time of cancer diagnosis Sex Qualitative Sex of the patient as found in the clinical history Ultrasound Nodule Size Quantitative Measurement of the diameters of the thyroid tumor on physical examination in mm Multifocality Qualitative Determination if the nodule is single or multiple Location Qualitative Location of the nodule within the gland: right, left, isthmus, or multiple Echogenicity Qualitative Determination of the echographic relationship with the rest of the thyroid parenchyma: very hypoechoic, hypoechoic, isoechoic, hyperechoic Composition Qualitative Ultrasound determination of whether the nodule is solid, predominantly solid, predominantly cystic, cystic, or spongiform Margins Qualitative Characterization of the nodule margins: smooth, irregular, lobulated, poorly defined, halo, extra-thyroidal extension Echogenic Foci Qualitative Presence of microcalcifications on ultrasound found within the nodule Shape Qualitative Nodule's greater dimension in height compared to its width on the transverse position of the transducer (taller-than-wide) TIRADS Quantitative Final suspicion value considering the parameters of each ultrasound, with values from I to V Bethesda Pathology Qualitative Classification according to Bethesda Follow-up Surgery Date Date of surgery if performed Date of First Examination Date of initial evaluation and start of surveillance Date of Last Control Date of the last known follow-up Reason for Surgery Qualitative Clinical or individual cause that led to the decision of surgery as treatment: growth, increased ultrasound suspicion, surgeon's decision, others Status at Last Control Qualitative Patient's condition at the last known evaluation: under surveillance or operated Type of Surgery Qualitative Type of surgery performed: hemithyroidectomy or total thyroidectomy Surveillance Time without Intervention Quantitative Time elapsed from the start of follow-up until surgery Final Surgical Pathology Qualitative/Quantitative Type of pathology result after examining the specimen post-surgery: benign, malignant, diagnostic Nodule Size Quantitative Measurement of the thyroid tumor diameters on physical examination in mm at the last ultrasound Size Variation Qualitative Size analysis compared to the initial: growth, decrease, or stable Increased Suspicion Qualitative Changes in ultrasound characteristics that increase suspicion of malignancy: high, intermediate, low, very low risk; ATA 2015 criteria Follow-up Time Quantitative Time of surveillance and follow-up in months without surgery after established surveillance 7. Ethical Considerations This research is classified as a no-risk study according to the guidelines of Resolution 008430 of 1993 for research involving human subjects, Article 11, Chapter I, Title II of the Ministry of Health of Colombia. Additionally, confidentiality of information is ensured, and during the study, ethical principles are respected. To guarantee confidentiality, each participant will be assigned a numerical code known only to the researchers.

11. Timeline The work is expected to be completed starting from the date of approval.

1. Months 1 to 8: Review of medical records, data collection
2. Months 8 to 12: Data analysis, writing of the final report

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thyroid nodules and FNAC with a report corresponding to Bethesda category IV-VI, treated at the following health centers: HUSVF, HAMA, Center of Excellence in Head and Neck Diseases - CEXCA, Somer Clinic.
2. Patients classified as low-risk tumors (intrathyroidal, with no evidence of locoregional or distant metastasis).
3. Patients not subjected to thyroidectomy as the initial treatment.

Exclusion Criteria:

* 1. Patients with a second head and neck cancer. 2. Patients with clinical or imaging evidence of thyroid malignancy with lymph node or distant metastasis confirmed by pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid nodules who underwent FNAC with a Bethesda IV-VI report
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
surgery-free survival. | 24 months
  Time elapsed from the start of follow-up until surgery or last visit

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Sanabria, Study Director — Universidad de Antioquia
Locations (4):
- Colombia (4):
  - Hospital Alma Mater de Antoquia, Medellín, Antioquia
  - Hospital San Vicente Fundacion, Medellín, Antioquia
  - Universidad de Antioquia, Medellín
  - Clinica Somer, Rionegro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smulever A, Pitoia F. Active surveillance in papillary thyroid carcinoma: not easily accepted but possible in Latin America. Arch Endocrinol Metab. 2019 Sep 2;63(5):462-469. doi: 10.20945/2359-3997000000168. eCollection 2019. PMID 31482955
- [Background] Rosario PW, Mourao GF, Calsolari MR. Active Surveillance in Adults with Low-Risk Papillary Thyroid Microcarcinomas: A Prospective Study. Horm Metab Res. 2019 Nov;51(11):703-708. doi: 10.1055/a-1015-6684. Epub 2019 Nov 4. PMID 31683339
- [Background] Garcia-Lozano CA, Sanabria A. Preliminary Report of Active Surveillance as a Conservative Strategy for Bethesda IV Thyroid Nodules. Thyroid. 2023 Jan;33(1):126-128. doi: 10.1089/thy.2022.0296. Epub 2023 Jan 4. No abstract available. PMID 36254389
- [Background] Sanabria A. Active Surveillance in Thyroid Microcarcinoma in a Latin-American Cohort. JAMA Otolaryngol Head Neck Surg. 2018 Oct 1;144(10):947-948. doi: 10.1001/jamaoto.2018.1663. PMID 30178005
- [Background] Sanabria A. Experience with Active Surveillance of Thyroid Low-Risk Carcinoma in a Developing Country. Thyroid. 2020 Jul;30(7):985-991. doi: 10.1089/thy.2019.0522. Epub 2020 Feb 20. PMID 31950887
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Molinaro E, Campopiano MC, Pieruzzi L, Matrone A, Agate L, Bottici V, Viola D, Cappagli V, Valerio L, Giani C, Puleo L, Lorusso L, Piaggi P, Torregrossa L, Basolo F, Vitti P, Tuttle RM, Elisei R. Active Surveillance in Papillary Thyroid Microcarcinomas is Feasible and Safe: Experience at a Single Italian Center. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e172-80. doi: 10.1210/clinem/dgz113. PMID 31652318
- [Background] Koot A, Soares P, Robenshtok E, Locati LD, de la Fouchardiere C, Luster M, Bongiovanni M, Hermens R, Ottevanger P, Geenen F, Bartѐs B, Rimmele H, Durante C, Nieveen-van Dijkum E, Stalmeier P, Dedecjus M, Netea-Maier R. Position paper from the Endocrine Task Force of the European Organisation for Research and Treatment of Cancer (EORTC) on the management and shared decision making in patients with low-risk micro papillary thyroid carcinoma. Eur J Cancer. 2023 Jan;179:98-112. doi: 10.1016/j.ejca.2022.11.005. Epub 2022 Nov 15. PMID 36521335
- [Background] Sugitani I, Ito Y, Miyauchi A, Imai T, Suzuki S. Active Surveillance Versus Immediate Surgery: Questionnaire Survey on the Current Treatment Strategy for Adult Patients with Low-Risk Papillary Thyroid Microcarcinoma in Japan. Thyroid. 2019 Nov;29(11):1563-1571. doi: 10.1089/thy.2019.0211. Epub 2019 Sep 25. PMID 31441377
- [Background] Brito JP, Ito Y, Miyauchi A, Tuttle RM. A Clinical Framework to Facilitate Risk Stratification When Considering an Active Surveillance Alternative to Immediate Biopsy and Surgery in Papillary Microcarcinoma. Thyroid. 2016 Jan;26(1):144-9. doi: 10.1089/thy.2015.0178. Epub 2015 Nov 5. PMID 26414743
- [Background] Tuttle RM, Fagin JA, Minkowitz G, Wong RJ, Roman B, Patel S, Untch B, Ganly I, Shaha AR, Shah JP, Pace M, Li D, Bach A, Lin O, Whiting A, Ghossein R, Landa I, Sabra M, Boucai L, Fish S, Morris LGT. Natural History and Tumor Volume Kinetics of Papillary Thyroid Cancers During Active Surveillance. JAMA Otolaryngol Head Neck Surg. 2017 Oct 1;143(10):1015-1020. doi: 10.1001/jamaoto.2017.1442. PMID 28859191
- [Background] Ito Y, Miyauchi A, Kihara M, Higashiyama T, Kobayashi K, Miya A. Patient age is significantly related to the progression of papillary microcarcinoma of the thyroid under observation. Thyroid. 2014 Jan;24(1):27-34. doi: 10.1089/thy.2013.0367. Epub 2013 Nov 14. PMID 24001104